CLINICAL TRIAL: NCT01409538
Title: Brain Imaging and Pain: Analysis of Placebo Analgesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R01 AT001424-05A; R01AT001424-05 (NIH)
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Brain Imaging of Placebo Analgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Asymptomatic control participants receive Natural History and Placebo instructions in a within-subject design. There are no patients, or active agents in this study. It is not a Clinical Trial.
  Interventions: Other: Placebo Instructions
- Control condition (Active Comparator): The control condition represents a no-intervention, repeated baseline control, since the "active" intervention in this study is placebo.
  Interventions: Other: Control condition

INTERVENTIONS:
Other: Placebo Instructions — There is no intervention in this study. It is not a Clinical Trial. The study is an investigation of the neural basis of placebo analgesia.
  Arms: Placebo
Other: Control condition — This protocol represents an investigation of the neural mechanisms of placebo analgesia. As such, it does not represent the traditional clinical trial design. Instead the "active" intervention is a placebo, and the comparison condition is a no-intervention control.
  Arms: Control condition

SUMMARY:
This study examines the brain activation associated with placebo pain reduction.

DETAILED DESCRIPTION:
This study is a basic science study of the mechanisms of placebo analgesia in asymptomatic healthy individuals. Each participant receives a baseline pain testing session, followed by a conditioning paradigm that results in expectation of pain relief and conditioning. They then undergo functional magnetic resonance imaging during either placebo (conditioned analgesia) or baseline. To examine order effects and habituation, the participants also either undergo a repeated placebo or a repeated baseline. The primary dependent measures in the study are the fMRI determined regions of interest, in a network of brain areas associated with pain processing. The anticipated outcome of the study is the alteration of network connectivity between sensory, affective, evaluative areas of the brain associated with placebo.

Because this is not a traditional clinical trial, there are not traditional efficacy criteria, rather the outcomes are changes in brain function from manipulations of patient expectation and classical conditioning.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* english speaking

Exclusion Criteria:

* pain condition
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Brain Imaging Results | 2 weeks from baseline
  This outcomes represents the neural network underpinnings of the placebo analgesic response. It is the result of a network analysis using structural equation modeling of fMRI determined brain activations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Robinson, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Sevel LS, O'Shea AM, Letzen JE, Craggs JG, Price DD, Robinson ME. Effective connectivity predicts future placebo analgesic response: A dynamic causal modeling study of pain processing in healthy controls. Neuroimage. 2015 Apr 15;110:87-94. doi: 10.1016/j.neuroimage.2015.01.056. Epub 2015 Feb 3. PMID 25659463
- [Background] Robinson ME, Staud R, Price DD. Pain measurement and brain activity: will neuroimages replace pain ratings? J Pain. 2013 Apr;14(4):323-7. doi: 10.1016/j.jpain.2012.05.007. PMID 23548484
- [Background] Letzen JE, Sevel LS, Gay CW, O'Shea AM, Craggs JG, Price DD, Robinson ME. Test-retest reliability of pain-related brain activity in healthy controls undergoing experimental thermal pain. J Pain. 2014 Oct;15(10):1008-14. doi: 10.1016/j.jpain.2014.06.011. Epub 2014 Jul 3. PMID 24998897
- [Background] Letzen JE, Craggs JG, Perlstein WM, Price DD, Robinson ME. Functional connectivity of the default mode network and its association with pain networks in irritable bowel patients assessed via lidocaine treatment. J Pain. 2013 Oct;14(10):1077-87. doi: 10.1016/j.jpain.2013.04.003. Epub 2013 Jun 3. PMID 23743257
- [Background] Kisaalita NR, Robinson ME. Analgesic placebo treatment perceptions: acceptability, efficacy, and knowledge. J Pain. 2012 Sep;13(9):891-900. doi: 10.1016/j.jpain.2012.06.003. Epub 2012 Jul 31. PMID 22854011
- [Background] Kisaalita N, Staud R, Hurley R, Robinson M. Placebo use in pain management: The role of medical context, treatment efficacy, and deception in determining placebo acceptability. Pain. 2014 Dec;155(12):2638-2645. doi: 10.1016/j.pain.2014.09.029. Epub 2014 Sep 28. PMID 25267208
- [Background] Craggs JG, Price DD, Robinson ME. Enhancing the placebo response: functional magnetic resonance imaging evidence of memory and semantic processing in placebo analgesia. J Pain. 2014 Apr;15(4):435-46. doi: 10.1016/j.jpain.2013.12.009. Epub 2014 Jan 9. PMID 24412799